CLINICAL TRIAL: NCT01850758
Title: A Randomized Controlled Trial of Regenexx™ SD Versus Exercise Therapy for Treatment of Partial and Complete, Non-retracted Anterior Cruciate Ligament Tears
Brief Title: Regenexx™ SD Versus Exercise Therapy for ACL Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regenexx, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RSI2013-RCT01
Record Dates: First submitted 2013-05-07; First posted 2013-05-09 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Anterior Cruciate Ligament Tear
Keywords: ACL; Anterior Cruciate Ligament; ACL Tear; Anterior Cruciate Ligament Tear; Partial ACL Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regenexx SD (Active Comparator): Bone Marrow Aspirate Concentrate injected under imaging guidance into the area of the damaged ligament.
  Interventions: Procedure: Regenexx SD
- Exercise Therapy (Active Comparator): Subjects will be instructed in a set of appropriate knee strengthening exercises and given an instructional hand-out to take home.
  Interventions: Other: Exercise Therapy

INTERVENTIONS:
Procedure: Regenexx SD — stem cell treatment
  Arms: Regenexx SD
Other: Exercise Therapy — exercise therapy control
  Arms: Exercise Therapy

SUMMARY:
The primary objective of this study is to compare the improvement in subject-reported clinical outcomes for Regenexx SD vs. Exercise Therapy treatment of partial and complete, non-retracted knee ACL ligament tears, from baseline to 3 months, with continued evaluation of efficacy and durability up to 24 months.

Secondary objectives include evaluation of MRI evidence of tendon repair; incidence of post-operative complications, adverse events, re-injections, and surgical intervention; change in pain score and use of pain medications.

DETAILED DESCRIPTION:
Prospective, randomized, controlled to include 25 subjects treated with Regenexx SD and 25 subjects treated with exercise therapy alone with the exercise group crossing over to the injection group at 3 months.

Subjects will have a partial or complete, non-retracted ACL ligament tear as evidenced with MRI.

Subjects will be enrolled within 60 days prior to Regenexx-SD injection or initiation of exercise therapy and take part in follow-up visits for two years following treatment. A preoperative visit will occur at the time of enrollment; follow-up visits will occur at the clinical site at 6 weeks, 3 months, 6 months, 12 months, and 24 months post injection.

The primary endpoint analysis will be conducted once all subjects reach the 3 month endpoint. Subjects will continue to be followed through the 2 year endpoint with data analysis performed at the 1 year and 2 year time points.

ELIGIBILITY:
Inclusion Criteria:

* Pain, swelling, or functional disability in the affected knee with activity, having failed conservative treatment (e.g. NSAIDs, physician initiated physical therapy) for at least 3 months or unable to return to normal day to day activities by 6 weeks
* Physical examination consistent with lax ACL ligament (Anterior Drawer Test)
* Abnormal Telos Arthrometer measurement
* Positive diagnostic MR imaging of the affected knee with at least 1/3 of the ACL ligament at any area along its length having high signal on MRI PDFS/Fat Sat images.
* Full range of motion of the affected knee (other than restriction clearly due to effusion)
* Normal range of motion of the non-treated knee
* Is independent, ambulatory, and can comply with all post-operative evaluations and visits

Exclusion Criteria:

* A massive ACL tear or one that includes more than 2/3'rds of the ligament that's retracted.
* Previous surgery to the affected ACL (i.e. previous ACL replacement with an autograft or allograft)
* Prior ACL prolotherapy, PRP, corticosteroid injection or other injection therapy within the past three months,
* Concomitant meniscus tear or cartilage injury that occurred at the same time as the as the ACL tear and which is considered a pain generator by the treating physician at the time intake into the study (i.e. a meniscus tear or cartilage lesion associated with an active BML).
* Concomitant PCL or LCL tears
* Inflammatory or auto-immune based joint diseases or other lower extremity pathology (e.g., rheumatoid arthritis, systemic lupus erythematosus, psoriatic arthritis, polymyalgia, polymyositis, gout pseudogout)
* Quinolone or Statin induced myopathy/ tendinopathy
* Kellgren-Lawrence grade 2 or greater knee osteoarthritis
* Significant knee extension lag compared to the opposite knee
* Symptomatic lumbar spine pathology (e.g. radicular pain)
* Severe neurogenic inflammation of the cutaneous nerves about the knee or thigh
* Contraindications for MRI
* Tested positive or has been treated for a malignancy in the past or is suspected of having a malignancy or is currently undergoing radiation or chemotherapy treatment for a malignancy anywhere in the body, whether adjacent to or distant from the proposed injection site
* Condition represents a worker's compensation case
* Currently involved in a health-related litigation procedure
* Is pregnant
* Bleeding disorders
* Currently taking anticoagulant or immunosuppressive medication
* Allergy or intolerance to study medication
* Use of chronic opioid,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05; Primary Completion 2020-05-22 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
IKDC Subjective Knee Evaluation Score Change from Baseline | Change from Baseline to 3 months
  The primary endpoint for this study is the difference between treatment groups in the within patient mean change from baseline to 3 months in IKDC scores.

SECONDARY OUTCOMES:
Mean Pain Scales | 3, 6, 12 and 24 months
  Difference between treatment groups in mean 0-10 pain scales at each follow-up timepoint
Magnetic Resonance Evaluation of ligament repair | 6 months
  Comparison of Magnetic Resonance Evaluation of ligament repair at 6 months
Mean IKDC Subjective Knee Evaluation Scores | 6, 12 and 24 months
  Difference between treatment groups in mean KDC Subjective Knee Evaluation Scores at 6, 12 and 24 months.
Incidence of complications and adverse events | 24 months
  Incidence and time to resolution of post-operative complications and adverse events between treatment groups.
Incidence of re-injection and surgical revision | 24 months
  Incidence of and time to re-injection and surgical revision between treatment groups.
Use of pain medications | 3, 6, 12 and 24 months
  Difference between treatment groups in use of pain medications at each follow-up timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Centeno, MD, Principal Investigator — Centeno-Schultz Clinic
Locations (1):
- Centeno-Schultz Clinic, Broomfield, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Centeno CJ, Berger DR, Pitts J, Markle J, Pelle AJ, Murphy M, Dodson E. Non-surgical treatment of anterior cruciate ligament tears with percutaneous bone marrow concentrate and platelet products versus exercise therapy: a randomized-controlled, crossover trial with 2-year follow-up. BMC Musculoskelet Disord. 2025 Sep 30;26(1):882. doi: 10.1186/s12891-025-09153-2. PMID 41029301